CLINICAL TRIAL: NCT04498338
Title: Effects of Neural Mobilization Augmented by Traditional Physical Therapy on Pain, Functional Disability and H-reflex in Patients After Lumbar Laminectomy: a Randomized Controlled Trial
Brief Title: Neural Mobilization and Conventional Physical Therapy After Laminectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Moussa Abdelfattah Youssif Sharaf, Assistant Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Interventional
Record Dates: First submitted 2020-07-29; First posted 2020-08-04 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Laminectomy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neural mobilization and conventional physical therapy (Experimental): Neural mobilization combined with conventional physical therapy program (Transcutaneous electrical nerve stimulation (TENs) and exercise program) were performed three times/week for 6 successive weeks.
  Interventions: Other: Neural mobilization combined with conventional physical therapy program
- Conventional physical therapy program (Active Comparator): Conventional physical therapy program (Transcutaneous electrical nerve stimulation (TENs) and exercise program) was performed three times/week for 6 successive weeks.
  Interventions: Other: Conventional physical therapy program

INTERVENTIONS:
Other: Neural mobilization combined with conventional physical therapy program — Neural mobilization of sciatic nerve combined with TENs and exercise program applied 3 times/week for successive 6 weeks.
  Arms: Neural mobilization and conventional physical therapy
Other: Conventional physical therapy program — TENs and exercise program applied 3 times/week for successive 6 weeks.
  Arms: Conventional physical therapy program

SUMMARY:
This study was conducted to evaluate the effect of addition of neural mobilization to a standard post-operative physical therapy program in patients with lumbar laminectomy.

DETAILED DESCRIPTION:
After Laminectomy, patients are suffering from many problems as pain, weakness. This study was conducted on two groups of patients who underwent lumbar Laminectomy as a surgical treatment for lumbar canal stenosis. The control group received TENS and strengthening exercises, while the study group received neural mobilization in addition to the program that was given to the control group. The outcome measures include pain intensity, nerve root compression and functional level which were measured pre-treatment and post-treatment through using visual analogue scale, H-reflex latency and Oswestry Disability Index (ODI) respectively.

ELIGIBILITY:
Inclusion Criteria:

* Aged from 35-50 years.
* Underwent lumbar laminectomy of one or two levels.

Exclusion Criteria:

* Patients who had arthritis in the joints of the lower limbs (which would limit walking).
* Patients who had tumors, fractures or infections of the spine.
* Patients who had diabetes mellitus.
* Patients who had polyneuropathy.
* Patients who had evidence of spinal cord compression.
* Patients who had previous spinal surgery.
* Patients who had spinal stability problems (e.g. spondilo-listhesis, spondilolysis).
* Patients who had sensory loss.

Ages: 35 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-03-31 (Actual); Primary Completion 2020-02-27 (Actual); Study Completion 2020-02-27 (Actual)

PRIMARY OUTCOMES:
Pain intensity | Up to 6 weeks
  It was evaluated through visual analogue scale (VAS). Visual analogue scale (VAS) is a 10-cm line with a "0" at the left end for "no pain" and 10 at the right end for "worst possible pain", each patient was asked to indicate on the line where his pain is in relation to the two extremes by circling the number.
Nerve root compression | Up to 6 weeks
  It was assessed through assessment of latency of H-reflex of S1. The participant was in prone-lying position. The active recording electrode was located on the soleus between the two heads of the gastrocnemius, while reference recording electrode was located on the Achilles tendon. The stimulation was applied at the midline in the popliteal fossa on the tibial nerve.

SECONDARY OUTCOMES:
Functional ability | Up to 6 weeks
  The functional ability was evaluated by Oswestery disability index (ODI). Oswestery disability index (ODI) is a valid and reliable tool for assessment of functional ability.
  The minimum value of this scale is 0. The maximum value of this scale is 100. The higher scores mean worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Moussa A Sharaf, Assist Prof, Principal Investigator — Cairo University, Egypt; Khalid Z Fouda, Assist Prof, Study Director — Cairo University, Egypt
Locations (1):
- Cairo University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-19): https://cdn.clinicaltrials.gov/large-docs/38/NCT04498338/Prot_SAP_000.pdf